CLINICAL TRIAL: NCT02523274
Title: Resveratrol and Exercise to Treat Functional Limitations in Late Life
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201500598 -N; R21AG049974 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Aging
MeSH Terms: interventions — Resveratrol; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo + exercise (Placebo Comparator): Placebo capsules will be taken orally daily in combination with exercise
  Interventions: Drug: Placebo; Behavioral: Exercise
- Resveratrol 500 mg/day + exercise (Experimental): 500 mg/day resveratrol taken orally in combination with exercise
  Interventions: Drug: Resveratrol; Behavioral: Exercise
- Resveratrol 1000 mg/day + exercise (Experimental): 1000 mg/day resveratrol taken orally in combination with exercise
  Interventions: Drug: Resveratrol; Behavioral: Exercise

INTERVENTIONS:
Drug: Resveratrol — Dietary compound commonly found in grapes and red wine. Will be given in 250 mg/day and 1000 mg/day dosages
  Arms: Resveratrol 1000 mg/day + exercise; Resveratrol 500 mg/day + exercise
Drug: Placebo — Vegetable-based cellulose
  Arms: Placebo + exercise
Behavioral: Exercise — Multi-modal exercise regimen, 3 days/week

SUMMARY:
The purpose of this research study is to evaluate the effects of combining physical exercise with a resveratrol supplementation on the physical function of older adults.

DETAILED DESCRIPTION:
This investigation is a pilot study to investigate the potential of resveratrol, a commercially-available nutritional product, to enhance the efficacy of physical exercise in improving physical function among older adults with functional limitations. The overarching objective of this project is to evaluate the safety and efficacy of an intervention combining resveratrol supplementation and physical exercise among sedentary persons aged > 65 years objectively-measured functional impairments. A total of 60 participants will be recruited to participate in this three month intervention study. All participants will engage in a center-based exercise program 3/days per week and will be randomly assigned to consume 1) placebo, 2) 500 mg/day resveratrol, or 3) 1000 mg/day resveratrol. This study will provide critical information regarding the influence of the combination of resveratrol and exercise on objectively-measured and self-assessed indices of physical function. The study will also provide novel biologic information regarding the relative effects of the interventions on skeletal muscle mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand study procedures and to comply with them for the entire length of the study
* Willingness to be randomized into either treatment group
* Age 65 years and older
* Physical limitations evidenced by >290 seconds needed to complete long-distance corridor walk test
* Sedentary lifestyle, defined as <150 min/wk of moderate physical activity as assessed by CHAMPS questionnaire

Exclusion Criteria:

* Failure to provide informed consent
* Regular consumption of a resveratrol supplement
* Current involvement in supervised rehabilitation program
* Absolute contraindication(s) to exercise training according to American College of Sports Medicine guidelines
* Pain classification > Grade 3 on Graded Chronic Pain Scale
* Peripheral vascular disease; peripheral neuropathy; retinopathy
* Severe cardiac disease, including:

NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina

* Myocardial infarction or stroke within past year
* Significant cognitive impairment, including:

known dementia diagnosis or a Mini-Mental State Examination exam score <24

* Progressive, degenerative neurologic disease (e.g., Parkinson's Disease, multiple sclerosis, ALS)
* Severe rheumatologic or orthopedic diseases (e.g., awaiting joint replacement, active inflammatory disease)
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 mos.
* Other significant co-morbid conditions that would impair ability to participate in the exercise-based intervention
* Simultaneous participation in another intervention trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buford, PhD, Principal Investigator — University of Alabama at Birmingham; Stephen Anton, Principal Investigator — University of Florida
Locations (1):
- UAB Center for Exercise Medicine, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo capsules will be taken orally following each meal three times daily
  Placebo: Vegetable-based cellulose
- Resveratrol 500 mg/Day: 500 mg/day resveratrol taken orally via capsule following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 500 mg/day and 1000 mg/day dosages
- Resveratrol 1000 mg/Day: 1000 mg/day resveratrol taken orally via capsule following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 500 mg/day and 1000 mg/day dosages
Period: Overall Study
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Started | 20 | 20 | 20
Completed | 19 | 18 | 18
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Resveratrol 500 mg/Day: 500 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 1000 mg/day and 1500 mg/day dosages
- Resveratrol 1000 mg/Day: 1000 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 1000 mg/day and 1500 mg/day dosages
- Total: Total of all reporting groups
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.72 (5.94) | 73.4 (5.63) | 73.8 (5.73) | 74.1 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 18 | 45
  Male | 6 | 7 | 2 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 14 | 13 | 16 | 43
  Non-Hispanic Black | 4 | 6 | 3 | 13
  Non-Hispanic other | 1 | 0 | 0 | 1
  Hispanic | 1 | 1 | 1 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (5.5) | 31.3 (7.6) | 32 (6.9) | 31.5 (6.7)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 98.4 (26.1) | 105 (20.3) | 103 (17.1) | 102.1 (21.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 140 (13.7) | 145 (15.1) | 133 (9.6) | 139.3 (12.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79.3 (11.8) | 82.4 (9.5) | 78.2 (8.2) | 80.0 (9.8)
Six-minute walk test [Mean (Standard Deviation); unit: m/s] | 1.0 (0.02) | 1.0 (0.02) | 1.0 (0.02) | 1.0 (0.02)
SPPB Total Score [Mean (Standard Deviation); unit: units on a scale] — Score on scale of 0-12. Higher score (closer to 12) indicates better functioning. Lower score (closer to 0) indicates lower functioning.
  units on a scale | 10.3 (0.2) | 10.4 (0.2) | 10.3 (0.2) | 10.3 (0.2)
Peak Knee Torque [Mean (Standard Deviation); unit: Newtons-Meter] — Peak knee torque measured by knee extension.
  Newtons-Meter | 73.3 (2.7) | 73 (2.6) | 71.7 (2.8) | 72.7 (2.7)
Late-Life Function and Disability Instrument [Mean (Standard Deviation); unit: Scores on a scale] — Method of assessing functional capacity and disability. Lower values correlate with lower functioning and higher values correlate with higher functioning.
  Scores on a scale | 73.6 (1.7) | 73.8 (1.7) | 73.6 (1.8) | 73.7 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed
Description: Walking speed is assessed by asking the participants to walk at their usual pace over a 4 m course. Participants are to stand with both feet touching the starting line and to start walking after a verbal command is given, and the time needed to complete the entire distance will be recorded. The faster of two walks will be used and changes between the groups at baseline and 12 weeks will be assessed.
Time Frame: Change at Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: m/s
Groups:
- Resveratrol 500 mg/Day: 500 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 500 mg/day and 1000 mg/day dosages
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Number analyzed (Participants) | 19 | 18 | 18
m/s | -0.04 [-0.1 to 0.03] | -0.03 [-0.09 to 0.04] | 0.04 [-0.02 to 0.11]

2. Secondary Outcome: Short Physical Performance Battery (SPPB).
Description: Investigators will assess lower-extremity function by asking the participants to perform a series of tasks including: walking at their usual pace over a 4 m course, repeated chair stands, and a balance test. Each task is scored from 0 to 4, with 4 indicating best level of performance and 0 the inability to complete the test. A summary score (0-12) is then calculated. Higher score on the scale is reflective of higher function and lower score reflects lower functioning. Changes between the groups at baseline and 12 weeks will be assessed.
Time Frame: Change between baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Resveratrol 500 mg/Day: 500 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 500 mg/day and 1500 mg/day dosages
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Number analyzed (Participants) | 19 | 18 | 18
score on a scale | 0.38 [-0.17 to 0.93] | 0.25 [-0.3 to 0.8] | 0.13 [-0.42 to 0.69]

3. Secondary Outcome: Isokinetic Strength.
Description: Isokinetic strength of the dominant limb will be assessed by a standard dynamometer and changes between the groups at baseline and 12 weeks will be assessed.
Time Frame: Change between baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Newtons-Meters
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Number analyzed (Participants) | 19 | 18 | 18
Newtons-Meters | -3.24 [-9.7 to 3.23] | 10.5 [4.28 to 16.7] | 6.15 [-0.31 to 12.6]

4. Secondary Outcome: 6-minute Walk Test
Description: Investigators will assess exercise capacity of participants using the six-minute (6-min) walk test to assess change in meters walked between the groups at baseline and 12 weeks.
Time Frame: Change between Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Number analyzed (Participants) | 19 | 18 | 18
Meters | 9.34 [-9.02 to 27.7] | 22.9 [4.18 to 41.6] | 33.1 [13.8 to 52.4]

5. Secondary Outcome: Late-Life Function and Disability Instrument
Description: The instrument includes 16 tasks representing a broad range of disability indicators that assesses both frequency of doing a task and perceived limitation. The instrument uses a scale from 0 to 100, with higher scores indicating higher levels of function.
Time Frame: Change at Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Resveratrol 500 mg/Day: 1000 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 1000 mg/day and 1500 mg/day dosages
- Resveratrol 1000 mg/Day: 1500 mg/day resveratrol taken orally following each meal three times daily
  Resveratrol: Dietary compound commonly found in grapes and red wine. Will be given in 1000 mg/day and 1500 mg/day dosages
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
Number analyzed (Participants) | 19 | 18 | 18
Score on a scale | 4.77 [0.06 to 9.49] | 5.72 [0.93 to 10.5] | 3.36 [-1.5 to 8.22]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Resveratrol 500 mg/Day | Resveratrol 1000 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 3/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Resveratrol 500 mg/Day (N=20) | Resveratrol 1000 mg/Day (N=20)
Heart Attack (Cardiac disorders) | 1 (20) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Resveratrol 500 mg/Day (N=20) | Resveratrol 1000 mg/Day (N=20)
Gastrointestinal Issues (Gastrointestinal disorders) | 3 | 2 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blood Sugar (Renal and urinary disorders) | 0 | 0 | 1
Bladder Infection (Hepatobiliary disorders) | 0 | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Elevated Blood Pressure (Vascular disorders) | 0 | 0 | 1
Heart Attack (Cardiac disorders) | 1 | 0 | 0
Light headedness (General disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02523274/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02523274/ICF_001.pdf